CLINICAL TRIAL: NCT00005722
Title: Stroke Belt Initiative
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4931
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Accident; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Hypertension

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
For State Health Departments located in Stroke Belt states, to assess high risk target audiences' needs and identify opportunities for more effective delivery of medical and/or educational services to reduce the high rate of stroke mortality experienced in the southeastern United States.

DETAILED DESCRIPTION:
BACKGROUND:

High blood pressure has long been established as the key risk factor for stroke, the third leading cause of death in the United States and a significant risk factor for coronary heart disease deaths. Cigarette smoking and obesity have also been found to be risk factors for stroke as well as heart disease.

Death rates from stroke differ by state. In 1980, eleven states had age-adjusted stroke mortality rates that were more than 10 percent higher than the United States average, 40.3 per 100,000. Ten of these eleven states (all except Indiana) were in the South, forming a "Stroke Belt". Florida's northern counties experienced higher stroke mortality rates than its southern counties, offering an opportunity for a comparative study.

In 1980, with few exceptions, each race/sex specific stroke death rate in the Stroke Belt states was more than 10 percent above the national average. Nonwhite men and women in the Stroke Belt had substantially higher rates than whites in the Stroke Belt and nonwhites elsewhere in the United States. However, whites in Stroke Belt states also had greater age-adjusted stroke death rates than did whites in other parts of the country.

In 1990, the National High Blood Pressure Education Program (NHBPEP) issued a Request for Proposals for the Stroke Belt Initiative. State Health Departments located in states with age-adjusted stroke mortality rates in excess of 10 percent of the national average were encouraged to initiate projects that assessed high risk target audience needs and to identify opportunities for more effective delivery of medical and/or educational services to reduce the high rate of stroke mortality experienced in the southeastern United States. These states were Alabama, Arkansas, Georgia, Indiana, Kentucky, Louisiana, Mississippi, North Carolina, South Carolina, Tennessee, and Virginia. In addition, the State of Florida was of interest because of differences in county age-adjusted stroke mortality rates--northern counties in the state experienced mortality rates as high or higher than rates in the Stroke Belt states, whereas southern counties exhibited rates closer to the national average, representing an excellent opportunity for a comparative study.

DESIGN NARRATIVE:

The Stroke Belt Initiative had two phases. In Phase I, the pilot phase, State Health Departments located in Stroke Belt states assessed high risk target audiences' needs and identified opportunities for more effective delivery of medical and/or educational services to reduce the high rate of stroke mortality experienced in the southeastern United States. This phase lasted for three years, from September 1990 through August 1993.

In the second phase, the State Health Departments used the methods and materials developed in the pilot phase to deliver health education interventions to reduce the overall risk of stroke.

ELIGIBILITY:
No eligibility criteria

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Study Completion 1996-09

CONTACTS AND LOCATIONS:
Overall Officials: Charles Barrett; Janice Bowie; Jerry Brown; Wendell Cox; Wendall Cox; Larry Deeb; Seth Emont; Carol Forbes; Barbara Hager; Jacquelyn Houston; Shirley Kirkconnell; Connie Pearson; Ramona Schaeffer; Canetta Washingon; Frances Wheeler; Donald Williamson; Gary Zelizer